CLINICAL TRIAL: NCT03997968
Title: A Multi-Center, Open Label Phase 1/2 Study of CYT-0851 in Patients With Relapsed/Refractory B-Cell Malignancies and Advanced Solid Tumors
Brief Title: A Phase 1/2 Study of CYT-0851 in B-Cell Malignancies and Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cyteir Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYT-0851-01
Record Dates: First submitted 2019-06-24; First posted 2019-06-25 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Malignancy; Non-hodgkin Lymphoma; Multiple Myeloma; Breast Cancer; Ovarian Cancer; Soft Tissue Sarcoma; Head and Neck Cancer; DLBCL; Mantle Cell Lymphoma; Follicular Lymphoma; Pancreatic Cancer; CLL; Small Cell Lung Cancer; Squamous Cell Carcinoma of Head and Neck; Triple Negative Breast Cancer
Keywords: Oral MCT-inhibitor; refractory; B-cell; solid tumor; cancer
MeSH Terms: conditions — Neoplasms; Lymphoma, Non-Hodgkin; Multiple Myeloma; Breast Neoplasms; Ovarian Neoplasms; Sarcoma; Head and Neck Neoplasms; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Pancreatic Neoplasms; Small Cell Lung Carcinoma; Squamous Cell Carcinoma of Head and Neck; Triple Negative Breast Neoplasms | interventions — Gemcitabine; Capecitabine; Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CYT-0851 dose escalation (Experimental): Part A: CYT-0851 administered orally in rising doses QD or BID for 28 day cycles
  Interventions: Drug: CYT-0851
- CYT-0851 dose expansion (Experimental): Part B: CYT-0851 administered orally at the selected Phase 2 dose for 28 day cycles
  Interventions: Drug: CYT-0851
- CYT-0851 and rituximab and bendamustine (Experimental): Part C: Daily oral doses of CYT-0851 for 28 days in combination with rituximab on Day 1 and bendamustine on Days 1 and 2 of each 28 day cycle
  Interventions: Drug: CYT-0851; Drug: CYT-0851 in combination with rituximab and bendamustine
- CYT-0851 and gemcitabine (Experimental): Part D: Daily oral doses of CYT-0851 for 28 days in combination with gemcitabine on Day 1, 8 and 15 of each 28 day cycle
  Interventions: Drug: CYT-0851; Drug: CYT-0851 in combination with gemcitabine
- CYT-0851 and capecitabine (Experimental): Part E: Daily oral doses of CYT-0851 for 21 days in combination with capecitabine on Days to 14 of each 21 day cycle
  Interventions: Drug: CYT-0851; Drug: CYT-0851 in combination with capecitabine

INTERVENTIONS:
Drug: CYT-0851 — Part A and B: Daily oral doses of CYT-0851 for 28 day cycles
Drug: CYT-0851 in combination with gemcitabine — Part D: Daily oral doses of CYT-0851 for 28 days in combination with gemcitabine
  Arms: CYT-0851 and gemcitabine
Drug: CYT-0851 in combination with capecitabine — Part E: Daily oral doses of CYT-0851 for 21 days in combination with capecitabine
  Arms: CYT-0851 and capecitabine
Drug: CYT-0851 in combination with rituximab and bendamustine — Part C: Daily oral doses of CYT-0851 for 28 days in combination with rituximab and bendamustine
  Arms: CYT-0851 and rituximab and bendamustine

SUMMARY:
This clinical trial is an interventional, active-treatment, open-label, multi-center, Phase 1/2 study. The study objectives are to assess the safety, tolerability and pharmacokinetics (PK) of CYT-0851 in patients with relapsed/refractory B-cell malignancies and advanced solid tumors and to identify a recommended Phase 2 dose as a monotherapy and in combination with chemotherapy for evaluation in these patients.

ELIGIBILITY:
Key Phase 1 Inclusion Criteria

1. Male or female ≥18 years of age at time of informed consent.

   1. Female subjects of childbearing potential must be non-lactating, not pregnant as confirmed by a negative serum pregnancy test at most 30 days before enrollment and within 72 hours before the first administration of CYT-0851
   2. Female subjects of childbearing potential must not donate ova during the study and for at least 90 days after the last dose of study drug and must agree to continue using an effective method of contraception during the screening period to first study drug administration until 90 days after the last dose of study drug
   3. Male subjects who have not had a vasectomy must agree to use an effective method of contraception during the study and until 90 days after the last dose of the study drug, and to not donate sperm during the study and for at least 90 days after the last dose of study drug
2. ECOG Performance Status of 0-1
3. Measurable disease defined by disease-specific response criteria
4. Histologically-proven B cell malignancies, meeting the following criteria:

   1. Relapsed, refractory B-cell non-Hodgkin lymphoma requiring therapy, after at least two prior therapies, and if transplanted, then at least 3-month post autologous stem cell transplant and if CART-treated, then evidence of progression no sooner than 3 months post CART treatment, or
   2. Relapsed, refractory chronic lymphocytic leukemia requiring therapy after at least two prior therapies, including BTK and BCL-2 inhibitor therapy (unless ineligible for such therapy), or
   3. For multiple myeloma, relapsed or progressive on or after treatment with at least three prior therapies that included a proteasome inhibitor, an imide, daratumumab, and if transplant eligible, a bone marrow transplant (unless unfit for transplant), or
5. Histologically-proven solid tumor meeting the following criteria:

   1. Patients must have failed, refused, or not be eligible for further standard therapies (including chemotherapy, hormonal therapies, Her-2 directed therapies, as appropriate) expected to provide clinical benefit, and meeting the following criteria
   2. Metastatic breast cancer (including ER/PR positive or negative, Her-2 positive and negative, triple negative), treated with at least 1 prior therapy for metastatic disease, or
   3. Recurrent squamous cell carcinoma of the head and neck (HNSCC) (dose escalation) or human papilloma virus positive (HPV+) HNSCC (dose-escalation and backfill), treated with at least 1 prior therapy, or
   4. Ovarian cancer, progressive after treatment with at least prior platinum-based chemotherapy, and therapy with a PARP inhibitor or
   5. Soft tissue sarcoma, treated with at least one line of prior systemic therapy, or
   6. Recurrent metastatic or locally advanced pancreatic cancer after first line chemotherapy (backfill or combination patients only) or
   7. Histologically-proven advanced small-cell lung cancer (SCLC) (monotherapy backfill patients only).

      1. Patients with mixed histology are not allowed
      2. Prior treatment with platinum containing chemotherapy regimen with no evidence of progression within 90 days of last dose of platinum agent and anti-PD-(L)1 unless contraindicated
      3. At least 1 prior line of chemotherapy, but no more than 3 prior lines of therapy
6. Understands the procedures and requirements of the study and provides written informed consent and authorization for protected health information disclosure
7. Willing and able to comply with the requirements of the study protocol
8. Site of disease amenable to a biopsy and willing to undergo biopsy required for backfill, or for dose-escalation if considered unsafe (approval to participate in the study required by the Medical Monitor) provide an archival sample ≤ 12 months old

Key Phase 2 Inclusion Criteria

1. Male or female ≥18 years of age at time of informed consent.

   1. Female subjects of childbearing potential must be non-lactating, not pregnant as confirmed by a negative serum pregnancy test at most 30 days before enrollment and within 72 hours before the first administration of CYT-0851
   2. Female subjects of childbearing potential must not donate ova during the study and for at least 90 days after the last dose of study drug and must agree to continue using, an effective method of contraception during the screening period to first study drug administration until 90 days after the last dose of study drug
   3. Male subjects who have not had a vasectomy must agree to use an effective method of contraception during the study and until 90 days after the last dose of the study drug, and to not donate sperm during the study and for at least 90 days after the last dose of study drug
2. ECOG Performance Status of 0-1
3. Measurable disease defined by disease-specific response criteria
4. Site of disease amenable to a biopsy and willing to undergo a biopsy for the determination of biomarker status, or, if considered unsafe (approval to participate in the study required by the Medical Monitor), archival sample ≤ 12 months old for determination of biomarker status.
5. Biomarker positive on recent biopsy or bone marrow sample if required for the specific cohort.
6. Histologically-proven B cell malignancies, meeting the following criteria:

   1. DLBCL Cohort

      1. Histologically-documented DLBCL or double hit lymphoma (B-cell lymphoma, unclassifiable, with features intermediate between diffuse large B-cell lymphoma and Burkitt lymphoma with BCL2 and MYC translocations (WHO Classification)
      2. Progressing on or after treatment with at least two prior lines of therapy, including R-CHOP or equivalent first line therapy
      3. If transplanted, then at least 3-month post autologous stem cell transplant
      4. If CART-treated, then evidence of progression no sooner than 3 months post CART treatment
   2. MCL Cohort

      1. Histologically-documented MCL
      2. Any stage at diagnosis
      3. Progressing on or after treatment with at least 2 prior lines of therapy, including a Bruton tyrosine kinase (BTK) inhibitor, after a 14-day washout period
   3. Multiple Myeloma Cohort

      1. Relapsed or progressing after treatment with at least 3 prior therapies that include a proteasome inhibitor, an Immunomodulatory imide drug (IMiD), daratumumab, and, if transplant eligible, a bone marrow transplant (unless unfit for transplant)
7. Or Histologically-proven solid tumors meeting the following criterial

   1. Patients must have failed, refused, or not be eligible for further standard therapies (including chemotherapy, hormonal therapies, Her-2 directed therapies, as appropriate) expected to provide clinical benefit, and meeting the following criteria
   2. Triple Negative Breast Cancer Cohort

      1. Histologically-documented triple negative breast cancer, ER/PR negative (defined as <10% of cells expressing hormonal receptors via immunohistochemistry (IHC) analysis), and HER2-negative, defined as either of the following by local laboratory assessment:

         * In situ hybridization (ISH) non-amplified (ratio of HER2 to CEP17 < 2.0 or single probe average HER2 gene copy number < 4 signals/cell), or
         * IHC 0 or IHC 1+
      2. At least 1 prior line of chemotherapy, but no more than 5 prior lines of chemotherapy
   3. Ovarian Cancer Cohort

      1. Histologically-proven metastatic epithelial ovarian cancer
      2. Prior treatment with a platinum containing chemotherapy regimen
      3. At least 1 prior line of therapy, but no more than 5 prior lines of chemotherapy
   4. Pancreatic Cancer Cohort

      1. Histologically-proven metastatic or locally advanced pancreatic cancer
      2. At least 1 prior line of chemotherapy but no more than 4 prior lines of systemic therapy
   5. Soft Tissue Sarcoma Cohort 1) Histologically-proven advanced soft-tissue sarcoma excluding all types of adipocytic sarcoma and GIST 2) At least 1 prior line of systemic therapy (unless no standard of care exists), but no more than 5 prior lines of systemic therapy
8. Follicular Lymphoma Cohort

   1. Histologically-documented follicular lymphoma
   2. Relapsed, refractory follicular lymphoma requiring therapy, after at least two prior therapies, and if CART-treated, then evidence of progression no sooner than 3 months post CART treatment
9. Understands the procedures and requirements of the study and provides written informed consent and authorization for protected health information disclosure
10. Willing and able to comply with the requirements of the study protocol

Key Exclusion Criteria

1. Medical Conditions

   1. Known history of HIV
   2. Known history of viral hepatitis B unless HBV viral load is below the limit of quantification and off viral suppressive therapy
   3. Know history of hepatitis C unless antiviral treatment with curative intent completed and HCV viral load is below the limit of quantification.
   4. Myocardial infarction or stroke within 6 months
   5. Uncontrolled hypertension (systolic blood pressure (SBP) > 160 or diastolic blood pressure (DBP) >100 on maximal medical therapy)
   6. History of interstitial pulmonary disease
   7. Unresolved pneumonitis
   8. Grade ≥ 3 neuropathy
   9. Known active central nervous system (CNS) metastases. Subjects with previously treated CNS metastases may participate as long as clinically and radiologically stable for at least 4 weeks after treatment, have no evidence of new or enlarging lesions and are off steroids and asymptomatic for 28 days prior to dosing with study medication
   10. Known history of meningeal involvement or meningeal carcinomatosis
   11. Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > 2 weeks prior to screening visit
   12. Presence of clinically significant cataracts
   13. Second malignancy, except treated basal cell or localized squamous skin carcinomas, localized prostate cancer, or other malignancy that is in remission or stable and for which patients have not been on active anti-cancer therapy for 2 years
   14. Pregnant or lactating. If β-HCG is elevated, eligible if ultrasound confirms absence of a pregnancy.
   15. Dementia or significantly altered metal status
   16. Bowel obstruction requiring medical management less than 4 weeks prior to screening
   17. Inability to tolerate oral intake that includes 2 full meals per day (or equivalent) or swallow pills.
   18. Recurrent ascites requiring paracentesis more frequently than every 4 weeks or within 14 days of screening.
   19. Weight loss of more than 10% over the preceding 3 months prior to screening
2. Prior/Concomitant Therapy

   1. Prior allogeneic stem cell transplant
   2. On systemic antibiotic, antifungal or anti-viral therapy
   3. White blood cell (WBC) growth factors administered within 14 days of screening visit
   4. Cancer therapy within 14 days prior to treatment with study drug
   5. On narrow therapeutic index medications that are sensitive substrates of CYP3A, P-gp or BCRP (or caution is warranted with approval by the Sponsor).
   6. On any drug known to prolong QTc interval (eg, certain antiarrhythmic, antimicrobials) that cannot be discontinued or interrupted 72 hours before the Day 1 dose through Day 2, and 72 hours before the Day 15 dose until Day 16 (BID dosing) or the Day 22 dose until Day 23 (QD dosing), in Cycle 1 (see Section 7.6.1 for a list of drugs).
   7. On systemic corticosteroid treatment for non-tumor indication at a daily dose equivalent to >10mg of Prednisone
3. Prior/Concurrent Clinical Study Experience a. Participation in another clinical trial (unless in the observation phase, or an observational study), or exposure to any investigational agent within 14 days prior to treatment with study drug
4. Laboratory assessments

   1. Complete blood count (CBC):

      Monotherapy and Chemotherapy Combinations 1 and 2:
      1. ANC < 1.0 × 10^9/L
      2. PLT < 75 × 10^9/L
      3. Hgb < 9.0 g/dL

         Chemotherapy Combination Group 3:

      1) ANC < 1.5 × 10^9/L 2) PLT < 100 × 10^9/L 3) Hgb < 9.0 g/dL

      Monotherapy and Chemotherapy Combination Groups 1 and 2:
   2. Calculated Creatinine clearance (Cockcroft-Gault) < 40 mL/min

Chemotherapy Combination Group 3:

b. Calculated Creatinine clearance (Cockcroft-Gault) < 50 mL/min c. Hepatic function

1. AST > 2.0 × ULN
2. ALT > 2.0 × ULN d. Total bilirubin > 1.5 x ULN e. Albumin < 2.8 g/dL 5. ECG Exclusion a. Screening QTc interval > 450 milliseconds for males and QTc > 470 ms for females (corrected by Fridericia) 6. Other Exclusions

   1. Unwilling or unable to make all planned study visits
   2. Unwilling or unable to provide a recent biopsy or bone marrow sample prior to enrollment and during study; Note: certain exceptions may be permitted allowing archival specimens prior to treatment or for subjects where a specimen is not required for biomarker positive testing
   3. Significant medical diseases or conditions, as assessed by the Investigators and Cyteir that would substantially increase the risk-benefit ratio of participating in the study. This includes but is not limited to acute myocardial infarction, arterial thrombosis, significant gastrointestinal bleed, or unstable angina within the last 6 months uncontrolled diabetes mellitus, current active infections, severely immunocompromised state, and congestive heart failure New York Heart Association (NYHA) Class III-IV, left ventricular ejection fraction (LVEF) < 40% d: Chemotherapy Combination Group 3 only: known history of dhydropyrimidine dehydrogenase deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Part A: Incidence of dose limiting toxicity | 28 Days
  Cycle 1 Dose limiting toxicities and determination of the maximum tolerated dose
Part B: Objective response rate | 24 Weeks
  clinical benefit as determined by investigator assessments of tumor response
Part C: Incidence of dose limiting toxicity | 28 Days
  Cycle 1 Dose limiting toxicities and determination of the maximum tolerated dose in combination with rituximab and bendamustine
Part D: Incidence of dose limiting toxicity | 28 Days
  Cycle 1 Dose limiting toxicities and determination of the maximum tolerated dose in combination with gemcitabine
Part E: Incidence of dose limiting toxicity | 21 Days
  Cycle 1 Dose limiting toxicities and determination of the maximum tolerated dose in combination with capecitabine

SECONDARY OUTCOMES:
Part A: Incidence of adverse events and other safety measures | 28 Days
  incidence of adverse events changes in laboratory parameters, vital signs and ECGs
  • Establish the PK of CYT-0851 Evaluate the type and frequency of adverse events
Part C: Incidence of adverse events and other safety measures | 28 Days
  incidence of adverse events changes in laboratory parameters, vital signs and ECGs
  • Establish the PK of CYT-0851 Evaluate the type and frequency of adverse events
Part D: Incidence of adverse events and other safety measures | 28 Days
  incidence of adverse events changes in laboratory parameters, vital signs and ECGs
  • Establish the PK of CYT-0851 Evaluate the type and frequency of adverse events
Part E: Incidence of adverse events and other safety measures | 21 Days
  incidence of adverse events changes in laboratory parameters, vital signs and ECGs
  • Establish the PK of CYT-0851 Evaluate the type and frequency of adverse events
Part A: Assessment of pharmacokinetic parameters | Phase 1: 12 months
  Summarize PK parameters including Cmax, AUC and tmax
Part C: Assessment of pharmacokinetic parameters | Phase 1: 12 months
  Summarize PK parameters including Cmax, AUC and tmax
Part D: Assessment of pharmacokinetic parameters | Phase 1: 12 months
  Summarize PK parameters including Cmax, AUC and tmax
Part E: Assessment of pharmacokinetic parameters | Phase 1: 12 months
  Summarize PK parameters including Cmax, AUC and tmax
Part B: Assessment of pharmacokinetic parameters | Phase 1: 12 months
  Summarize PK parameters including Cmax, AUC and tmax
Part A: Objective response rate | 24 months
  clinical activity as assessed by investigator assessment of objective response and duration of response
Part C: Objective response rate | 24 months
  clinical activity as assessed by investigator assessment of objective response and duration of response
Part D: Objective response rate | 24 months
  clinical activity as assessed by investigator assessment of objective response and duration of response
Part E: Objective response rate | 24 months
  clinical activity as assessed by investigator assessment of objective response and duration of response
Part B: Anti-tumor activity and by DOR | 24 months
  Antitumor activity as assessed by duration of response
Part B: Anti-tumor activity by PFS | 24 months
  Antitumor activity as assessed by progression free survival
Part B: Anti-tumor activity by DCR | 24 months
  Antitumor activity as assessed by disease control rate
Part B: Anti-tumor activity by OS | 24 months
  Antitumor activity as assessed by overall survival
Part B: Safety assessment | 24 months
  Safety as determined by incidence of AEs and SAEs and changes in laboratory, vitals and ECG findings

CONTACTS AND LOCATIONS:
Overall Officials: Markus Renschler, MD, Study Director — Cyteir Therapeutics
Locations (16):
- United States (16):
  - University of California San Francisco, San Francisco, California
  - Stanford Comprehensive Cancer Center, Stanford, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists and Research Institute, Sarasota, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - John Theurer Cancer Center at HUMC, Hackensack, New Jersey
  - NYU Langone Health, New York, New York
  - Oklahoma University-Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Washington Seattle Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No